CLINICAL TRIAL: NCT04939727
Title: Suicide Prediction and Prevention for People at Risk for Opioid Use Disorder: Supplement to COMPUTE 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A20-042; 3UG1DA040316-06S3 (NIH)
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-04

CONDITIONS: Opioid Use; Opioid-use Disorder; Suicide
Keywords: OUD; Opioid Use Disorder Treatment; Suicide prevention; Suicide risk
MeSH Terms: conditions — Opioid-Related Disorders; Suicide; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OUD-CDS + Suicide Risk Model associated CDS (Intervention arm) (Experimental): Providers that practice in the clinics in this intervention arm will receive access to the OUD-CDS + Suicide Risk Model associated CDS, for all eligible encounters.
  Interventions: Other: OUD-CDS + Suicide Risk Model associated CDS
- Control (No Intervention): Providers that practice in the clinics in this control arm will not receive any access to the OUD-CDS + Suicide Risk Model associated CDS, however these clinical decision-support tools will run "silently" in the background, collecting data on eligible encounters.

INTERVENTIONS:
Other: OUD-CDS + Suicide Risk Model associated CDS — Access to OUD-CDS + Suicide Risk CDS
  Other Names: Suicide Risk CDS
  Arms: OUD-CDS + Suicide Risk Model associated CDS (Intervention arm)

SUMMARY:
This study integrates the Mental Health Research Network (MHRN) suicide risk models into Opioid Wizard, an electronic health record (EHR) clinical decision support (CDS) to identify and treat patients at high risk of opioid use disorder (OUD)/overdose or diagnosed with OUD, to alert primary care clinicians (PCCs) to patients at elevated risk for suicide and guide them through structured suicide risk assessment. In both intervention and control clinics, suicide risk scores will be calculated for all Opioid Wizard-eligible patients and relevant EHR data to inform analyses will be archived. In intervention clinics, Opioid Wizard will alert PCCs to Opioid Wizard-eligible patients who are at increased risk of suicide and coach them through use of the Columbia Suicide Severity Risk Scale (CSSRS), a structured tool in the EHR that will help PCCs assess immediate suicide risk. Based on the resulting CSSRS score, Opioid Wizard will provide EHR links for risk-based referrals and follow-up recommendations, including care as usual, routine or emergent referral to behavioral health, or transportation to the emergency department (ED) for further assessment. Primary outcome measures include completion of CSSRS assessments for at-risk patients and patient engagement in outpatient mental health care.

DETAILED DESCRIPTION:
When a patient is at elevated risk of suicide, the PCC will be prompted by Opioid Wizard to complete the CSSRS, easily available to all PCCs in the EHR and saved as discrete data elements. Risk-based (depending on CSSRS score) referral and follow-up recommendations for suicide prevention will be given, with specific care recommendations ranging from care as usual (very low risk) to referral to behavioral health for evaluation and safety planning (moderate to high risk) to immediate evaluation in the emergency department and potential inpatient admission (very high risk), building on workflows developed for use by care managers in in our recently completed suicide prevention trial of over 19,000 people at elevated risk of suicide. (28) The MHRN suicide risk models will be programmed into the EHR, a rigorous process that will take approximately 6 months. This process includes building the model in a testing environment in the EHR, testing the model with fictitious patients in a EHR testing environment and conducting chart audits, revising as needed, testing the model in a different EHR testing environment with real patient data, revising as needed, testing the model by running it silently in the EHR production environment and conducting chart audits, and revising as needed. This is followed by testing in the EHR production environment with 5-15 physicians in 1-2 pilot clinics. Prior to the go-live date for the suicide risk calculator, training on use and interpretation of the suicide risk model and the CSSRS will be provided to all PCCs and their rooming staff in intervention clinics. Training for control clinics will be separate and will provide training on the use of the CSSRS.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18-75 years, inclusive, at the time of index visit
2. Have an OUD diagnosis, be prescribed an active MOUD, or be identified by the opioid risk models as being at high risk of OUD or overdose
3. Be identified at high risk of suicide by the suicide risk models

Exclusion Criteria:

1. Active parenteral chemotherapy within the last year
2. Stage 4 or equivalent cancer diagnoses
3. Enrolled in hospice or palliative care programs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Rossom, MD, MSCR, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute, Bloomington, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study patients had index visits at randomized clinics between August 3, 2021 and April 30, 2022. The index visit was the first visit during the accrual period at which the patient met all study eligibility criteria. First participant enrolled on August 3rd, 2021.
Units Other Than Participants: Primary Care Clinics
Period: Overall Study
Arm/Group | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) | Control
Started | 69; 8 Primary Care Clinics | 46; 7 Primary Care Clinics
Completed | 69; 8 Primary Care Clinics | 46; 7 Primary Care Clinics
Not Completed | 0; 0 Primary Care Clinics | 0; 0 Primary Care Clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) | Control | Total
Number analyzed (Participants) | 69 | 46 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.2) | 37.6 (12.0) | 39.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 27 | 65
  Male | 31 | 19 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 65 | 45 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 54 | 39 | 93
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 46 | 115
Medicaid [Count of Participants; unit: Participants] | 57 | 38 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With CSSRS Completion on the Same Day or in the 14 Days Following Any Outpatient Visit
Description: EHR documentation of a completed Columbia Suicide Severity Rating Scale (CSSRS) on the same day or in the 14 days following any outpatient visit during the observation period.
Time Frame: Observation period (up to 12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) | Control
Number analyzed (Participants) | 69 | 46
Participants | 14 | 8

2. Primary Outcome: Number of Outpatient Visits With Adequate Mental Health Engagement
Description: Adequacy of engagement with mental health care following outpatient visits that occurred between the index visit and the end of the study period. Engagement was adequate if acute suicide risk was 1) documented as moderate or high and the patient had a follow-up mental health visit within 30 days, or 2) undocumented but the patient had a follow-up mental health visit within 30 days, or 3) documented as low.
Time Frame: Observation period (up to 12 months)
Population: All outpatient visits between enrollment and the end of the observation period were assessed for appropriate outpatient mental health care engagement. Multiple visits per patient were possible during this time period.
Measure: Count of Units; unit: Outpatient visits
Units Other Than Participants: Outpatient visits
Arm/Group | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) | Control
Number analyzed (Participants) | 69 | 46
Number analyzed (Outpatient visits) | 911 | 554
Outpatient visits | 789 | 489

3. Primary Outcome: Number of Participants With One or More Suicide Attempts
Description: Identification of fatal or non-fatal suicide attempts, using ICD-10 diagnostic codes assigned at inpatient or outpatient visits during the outcome measure time frame
Time Frame: Two time periods: 1) 12 months prior to enrollment (index visit), and 2) between enrollment and end of observation period (up to 12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) | Control
Number analyzed (Participants) | 69 | 46
Participants
  12 months prior to enrollment | 19 | 15
  Between enrollment and observation period | 3 | 0

4. Primary Outcome: Number of Participants With One or More Opioid Overdoses
Description: Identification of opioid overdoses, using ICD-10 diagnostic codes assigned at inpatient or outpatient visits during the outcome measure time frame
Time Frame: Two time periods: 1) 12 months prior to enrollment (index date), and 2) between enrollment and end of observation period (up to 12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) | Control
Number analyzed (Participants) | 69 | 46
Participants
  12 months prior to enrollment | 8 | 7
  Between enrollment and end of observation period | 2 | 5

ADVERSE EVENTS:
Time Frame: Between enrollment (index date) and end of observation period (up to 12 months).
Arm/Group | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) | Control
All-Cause Mortality (participants affected / at risk) | 3/69 | 0/46
Serious Adverse Events (participants affected / at risk) | 46/69 | 23/46
Other Adverse Events (participants affected / at risk) | 6/69 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) (N=69) | Control (N=46)
Emergency Department Encounter (General disorders) | 42 | 22 — Emergency department encounter for any reason
Inpatient stay (General disorders) | 14 | 5 — Inpatient stay for any reason
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OUD-CDS + Suicide Risk Model Associated CDS (Intervention Arm) (N=69) | Control (N=46)
Overdose (General disorders) | 6 | 3 — Poisoning by or toxic affect of any agent

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT04939727/Prot_SAP_000.pdf